CLINICAL TRIAL: NCT02163148
Title: Predictors of Exposure Success in Public Speaking Anxiety
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tali Manber Ball, Doctoral Candidate, University of California, San Diego
Other Study IDs: UCSDIRB-130313
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Performance Anxiety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Public Speaking Anxiety: Intervention to be administered: One speech exposure session.
  Interventions: Behavioral: Massed speech exposure session

INTERVENTIONS:
Behavioral: Massed speech exposure session — One session consisting of 4 speech exposures, each 5 minutes long.

SUMMARY:
Anxiety disorders are common and impairing. Although exposure therapy is one of the most effective treatments for anxiety, some individuals do not fully respond to treatment, and these individual differences are not well understood. Exposure therapy involves repeated, deliberate, safe engagement with a feared stimulus without the feared outcome occurring. This treatment is thought to work through a type of emotional learning called fear extinction. This study aims to look at links between fear extinction learning and exposure success, with the overall goal of better understanding who is likely to respond best to exposure therapy and why.

ELIGIBILITY:
Inclusion Criteria:

* Score of at least 20 on the PRCS
* Age 18-55
* English fluency

Exclusion Criteria:

* Psychotropic medication use in the past 4 weeks
* Past experience with exposure based therapy
* History of bipolar disorder, psychotic disorder, or substance dependence
* Current major depressive disorder of greater than moderate severity (defined as a score on the 9 item Patient Health Questionnaire of greater than 14)
* Clinically significant suicidal or homicidal ideation
* Non-removable ferrous metal
* Current significant neurological conditions
* History of loss of consciousness greater than 5 minutes duration
* Pregnant
* Claustrophobic

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in peak Subjective Unit of Distress (SUDS) rating from first to fourth (last) exposure | 90 minutes
  Participants will complete 4 exposures during one 90 minute session. Change in the peak ratings on the final exposure relative to the first exposure will be the outcome measure.

SECONDARY OUTCOMES:
Change from baseline on the Liebowitz Social Anxiety Scale (LSAS) at 2 weeks | Baseline, week 2
Change from baseline on the Personal Report of Confidence as a Speaker (PRCS) at 2 weeks | Baseline, week 2

OTHER OUTCOMES:
Change from baseline on the Sheehan Disability Scale (SDS) at week 2 | Baseline, week 2

CONTACTS AND LOCATIONS:
Overall Officials: Tali M Ball, MA, Principal Investigator — UCSD
Locations (1):
- UCSD Psychiatry Research, San Diego, California, United States

REFERENCES:
- [Derived] Ball TM, Knapp SE, Paulus MP, Stein MB. Brain activation during fear extinction predicts exposure success. Depress Anxiety. 2017 Mar;34(3):257-266. doi: 10.1002/da.22583. Epub 2016 Dec 6. PMID 27921340